CLINICAL TRIAL: NCT00778297
Title: Immunogenicity and Tolerability Study of FluvalAB FL-K-004 Trivalent Influenza Vaccine With 6 Mcg HA/Strain/Dos Antigen Content
Brief Title: Immunogenicity and Tolerability Study of FluvalAB FL-K-004 Trivalent Influenza Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fluart Innovative Vaccine Ltd, Hungary (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FluvalAB-H-05; OGYI 28438/82/07; EudraCT 2007-004239-52
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Influenza
Keywords: prevention; influenza; infection; vaccine; Influenza vaccine; Influenza in humans
MeSH Terms: conditions — Influenza, Human; Infections | interventions — Vaccination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental)
  Interventions: Biological: Vaccination with FluvalAB FL-K-004 trivalent flu vaccine
- Group 2 (Active Comparator)
  Interventions: Biological: Vaccination with FluvalAB trivalent influenza vaccine

INTERVENTIONS:
Biological: Vaccination with FluvalAB FL-K-004 trivalent flu vaccine — Treatment: 6 μg HA/strain/dos of FluvalAB FL-K-004 trivalent influenza vaccine will be administered once (at Day 0).
  Arms: Group 1
Biological: Vaccination with FluvalAB trivalent influenza vaccine — Treatment: 15 μg HA/strain/dos of FluvalAB trivalent influenza vaccine will be administered once (at Day 0).
  Arms: Group 2

SUMMARY:
This is a single blind, reference drug controlled, one center viral immunogenicity and tolerability study of FluvalAB FL-K-004 Trivalent Influenza Vaccine with 6 μg HA/strain/dos antigen content to assess immunogenicity and tolerability.

The aim of the study is to assess the immunogenicity and tolerability of FluvalAB FL-K-004 trivalent influenza vaccine with 6 μg HA/strain/dos antigen content (study drug) in age groups 18-60 years and over 60 years, with the objective to verify efficacy and tolerability of the study drug according to CPMP/BWP/214/96: "Note for Guidance on Harmonization of Requirements for Influenza Vaccines", 12 March 1997.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers in good health aged over 18 years, both sexes;
* Full contractual capacity of the participants;
* Are in good health (as determined by vital signs and medical history);
* Negative urine or serum pregnancy test for females of childbearing potential;
* Are able to understand and comply with planned study procedures;
* Signed informed consent prior to initiation of study procedures;
* Absence of existence of any exclusion criteria.

Exclusion Criteria:

* Known allergy to eggs or other components of the vaccine;
* History of Guillain-Barré syndrome;
* Pregnancy or breast feeding or positive pregnancy test prior to vaccination;
* Immunosuppressive therapy in the preceding 36 months;
* Active neoplasm (i.e. requiring any form of anti-neoplastic therapy);
* Concomitant corticosteroid therapy, including inhaled corticosteroids;
* Psychiatric illness and/or concomitant psychiatric drug therapy;
* Immunoglobulin (or similar blood product) therapy within 3 months prior to vaccination;
* Vaccine therapy within 4 weeks prior to the study;
* Influenza vaccination within 6 months prior to the study;
* Chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the immune response;
* Documented HIV, HBV or HCV infection;
* Acute febrile respiratory illness within one week prior to vaccination;
* Experimental drug therapy within 1 month prior to vaccination;
* Alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Post-vaccination HI antibody titre | 21-28 days after vaccination
Incidence of adverse reactions | 21-28 days after vaccination

SECONDARY OUTCOMES:
Post-vaccination HI antibody titer | 110-120 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ferenc Tamás, MD, Principal Investigator — Pilisvörösvár District Doctor's Office; Zsuzsa Galambos, MD, Study Director — Omninvest Ltd.
Locations (1):
- Pilisvörösvár District Doctor's Office, Pilisvörösvár, Hungary